CLINICAL TRIAL: NCT05125783
Title: Multifactorial Analysis of the Influence of Alcohol Marketing Stimuli in Adults With Regular Alcohol Consumption on the Perception of Alcohol Risks and According to Types of Use and Individual Vulnerabilities
Brief Title: Influence of Alcohol Marketing Stimuli in Adults With Regular Alcohol Consumption
Acronym: DEPREV_Phase_2
Status: Terminated | Type: Observational
Why Stopped: Recruitment difficulties
Sponsor: University Hospital, Brest (Other)
Collaborators: Ecole des Hautes Etudes en Santé Publique (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0178
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-03

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Completion of the questionnaire by the patient after consultation with the practitioner.

SUMMARY:
Alcohol use is the second leading cause of preventable death after smoking. The Evin law was built in 1991 with the goal of reducing exposure to alcohol marketing among the youngest. But this law is currently extremely weakened, and in a press release of February 26, 2018, the French Society of Alcoology is alarmed by these developments.

Studies on the impact of alcohol marketing focus for the most part on young adolescents and the links between marketing exposure and alcohol initiation. But beyond these links, little work has been done on the impact of alcohol marketing on vulnerable subjects with regular alcohol consumption. Alcohol consumption is one of the very first causes of hospitalization in France. The damage is often limited to the notion of risks of dependence, but it can appear as soon as consumption of 1 standard unit/day and mainly concerns the 45-64 year olds. To investigator knowledge, there are no studies on the impact of alcohol marketing carried out among regular alcohol users with moderate or severe alcohol use disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient with moderate to severe alcohol use disorders (beyond 3 out of 11 criteria on the DSM-5 scale)
* Non-opposition of the patient

Exclusion Criteria:

* Minor patient
* Patient who has already participated in phase 1 of the project
* Non-comprehension of the written French language
* Refusal to participate in the study
* Patient of legal age, deprived of liberty by a judicial or administrative decision or unable to express their consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age followed in the addictology services participating in the study with moderate or severe alcohol use disorders.
Sampling Method: Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Alcohol marketing strategies | 1 day
  Confirmation of alcohol marketing strategies significantly influencing alcohol risk perception alcohol cravings in patients with moderate to severe alcohol use disordersin a large population of people with alcohol use disorders seeking care.

SECONDARY OUTCOMES:
Alcohol craving | 1 day
  Self-assessment of craving measured by a visual analog scale from 0 (no craving for alcohol) to 10 (irrepressible craving for alcohol) relative to the question "How much do you estimate your craving for alcohol? "
Alcohol consumption | Day 1
  Ability to control one's drinking, as measured by a visual analog scale from 0 (no ability to control) to 10 (perceived total control over drinking) relative to the question "How much do you estimate your ability to control your own drinking?"
Evaluation of severity of alcohol use disorders | Day 1
  Severity of alcohol use disorders as measured by the number of DSM5 (Diagnostic and Statistical manual of Mental disorders 5) criteria. The DSM5 score is diagnosis of addiction is based on welldefined criteria set out in the Diagnostic and Statistical manual of Mental disorders (DSM), the fifth edition of which was published in 2013. The questionnaire consists of 11 items (diagnostic criteria for substance use disorders from the American Psychiatric Association's DSM V). The presence of 2 to 3 criteria: low addiction / Presence of 4 to 5 criteria : moderate addiction / Presence of 6 or more criteria: severe addiction.
Evaluation of severity of alcohol use disorders | Day 1
  Severity of alcohol use disorders as measured will be evaluated by Alcohol Use Disorders Identification Test (AUDIT) scale. AUDIT is a 10-item screening tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems. A score of 8 or more is considered to indicate hazardous or harmful alcohol use.
Socio-demographic characteristics | Day 1
  The impact of marketing stimuli will be evaluated according to socio-demographic characteristics.
Alcohol consumption | Day1
  Assessment of the type of alcohol consumption

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Les Apsyades, Bouguenais
  - François-Néri VANDERMERSCH, Bouguenais
  - Morgane GUILLOU-LANDREAT, Brest
  - Jean-Pierre SIMSON, Brest
  - Pascale ROZEC, Landerneau
  - Benoit SCHRECK, Nantes
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement